CLINICAL TRIAL: NCT06547580
Title: Examining the Effects of Group-based and Individual Pelvic Floor Muscle Training on Elderly Individuals With Urinary Incontinence
Brief Title: Effects of Group-based and Individual Pelvic Floor Muscle Training on Elderly Individuals With Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CelalBayarU1
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence; pelvic floor muscle training; elderly people; elektromyography
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-based PFMT (Experimental): A group-based Pelvic floor muscle training was practiced under the supervision of an experienced physiotherapist, 2 sessions a week, 30-45 minutes each, for 12 weeks.
  Interventions: Other: Group-based PFMT
- Individualized PFMT (Experimental): Individualized Pelvic floor muscle training with Electromyography Biofeedback was practiced under the supervision of an experienced physiotherapist, 2 sessions a week, 30-45 minutes each, for 12 weeks.
  Interventions: Other: Individualized PFMT

INTERVENTIONS:
Other: Group-based PFMT — Under the supervision of an experienced physiotherapist, group-based pelvic floor muscle training was applied for 12 weeks, 2 sessions per week, 30-45 minutes each session.
  Arms: Group-based PFMT
Other: Individualized PFMT — Under the supervision of an experienced physiotherapist, individualized pelvic floor muscle training was performed using the Emg Biofeedback device, 2 sessions a week, 30-45 minutes each session, in 12 weeks.
  Arms: Individualized PFMT

SUMMARY:
The purpose of this study is to asses the effects of 12-week group-based and individually planned pelvic floor muscle training on individuals aged 65 and over with urinary incontinence.

DETAILED DESCRIPTION:
The research was conducted on participants over the age of 65 with urinary incontinence living in a nursing home. After these participants were informed about the content of the study, a signed informed consent form will be obtained. This study is an assessor-blinded, randomized controlled trial. Participants with incontinence aged 65 and over living in a nursig home were randomly assigned to intervention (IG) and control group (CG). The intervention group attended an exercise program that individualized pelvic floor muscle with Emg biofeedback training (individualized-PFMT). The control group was included in the group-based PFMT program. Duration of exercise for both groups was 45-60 minutes per session three times a week for 12 weeks. Incontinence symptoms and severity (Pelvic Floor Distress Inventory-20, bladder diary), PFM and abdominal muscle function (superficial electromyography), balance (Berg Balance Scale), functional status (Senior Fitness Test), hand grip strength, knee extansor, ankle dorsi-plantar flexion muscle srength, sleep quality and fear of falling (Falls Efficacy Scale) was measured at baseline and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Having signed the informed volunteer consent form
* Being 65 years or older
* Having urinary incontinence
* Ability to walk unaided and not use any walking aids

Exclusion Criteria:

* Having severe walking and balance problems
* Severe cognitive impairment (Mini mental state assessment test score below
* Having a serious neurological problem
* Having serious heart diseases
* Having a genito-urinary infection
* Having pelvic organ prolapse
* Six months ago he received medication for incontinence
* Having had incontinence and abdominal surgery
* Having metastatic cancer
* Having any vision problems

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
incontinence symptoms and severity | baseline and week 12 (after intervention)
  SPSS 29 is validated. Pelvic Floor Distress Inventory-20 (PFDI-20) instrument scores were recorded at the baseline and after the intervention. Pelvic Floor Distress Inventory-20 Scale evaluates pelvic organ prolapse, urinary and colorectoanal problems that may develop due to pelvic floor dysfunction, and the degree of complaints about them; It is the short form of the Pelvic Floor Distress Inventory Scale. While the best score for each subheading is 0 and the worst score is 100.
  Change: Week 12- baseline
balance | baseline and week 12 (after intervention)
  SPPS 29 is validated. Berg Balance Scale score will be recorded at baseline and after the intervention. It consists of fourteen items. The proficiency level in the activity for each item is 0; "cannot", 4; It is indicated with 5 points (0-4), "makes it independent and safe". The 14 functional parameters included in Berg Balance Scale. The maximum score that participants can get from the test is 56 and reflects an excellent balance function. (0-20 points; severe fall risk, 21-40 points; moderate fall risk, 41-56; mild fall risk). The fall risk limit for this test is 45 points.Change: Week 12- baseline
Bladdery diary | baseline and week 12 (after intervention)
  SPPS 29 is validated. The patient records the type and amount of fluid he/she takes, the frequency of urinary incontinence, the urination volume, the frequency of urination at night, and the situations in which he/she leaks urine, along with the times in a 24-hour voiding diary. It is an objective evaluation method used to determine the type and degree of incontinence.
  Change: Week 12- baseline.
Senior fitness test- functional performance-30-second chair stand test | baseline and week 12 (after intervention)
  SPPS 29 is validated. 30-second chair stand test score were recorded at the baseline and after the intervention.
  The participant was asked to sit in the middle part of a 43.18 cm (12in) high chair with his back upright, feet on the ground and arms crossed in front of his chest (right hand on the left shoulder, left hand on the right shoulder). While in this position, the participant starts the test with the start command and takes off as fully as he can during 30 seconds. The number of complete takes off during 30 seconds determines the score.A score of less than 10 in 30 seconds indicates lower extremity muscle weakness.
  Change: Week 12- baseline.
Senior fitness test- functional performance-Eight (2.45m) Food Up and Go Test | baseline and week 12 (after intervention)
  SPPS 29 is validated.For the test, which is used to evaluate functional mobility and dynamic balance in elderly participants, the participants was seated in a chair with a backrest and armrests, with his back and arms supported. After the command to "get up" was given to the patient, he was asked to walk at his normal speed to an object placed 2.45 m away from the chair, and then turn around the object and walk back. The period started when the patient was commanded to "get up" and was stopped when he/she sat on the chair.
  Change: Week 12- baseline.
Senior fitness test- functional performance-Chair Sit and Reach Test | baseline and week 12 (after intervention)
  SPSS 29 is validated.This test, is used especially to determine the flexibility of the hamstring muscle group. The participant was seated on a 43.18 cm high chair leaning against a wall or a solid place, with the junction of the thigh and hip bones in front of the chair. The participant was allowed to extend one foot forward, in full extension, with the heel on the ground and the ankle at approximately 90 degrees, leaving it to the participant's own choice (right or left). The participant was told to stretch his body forward with both hands, without bending his extended knee, and to reach towards his toe without pushing the pain limit. Participant; If the fingertips do not touch the tip of the foot, the distance between them, in centimeters (-), is the participant's; If the fingertips of the middle hand touch the tip of the foot, zero (0) is given to the participant.
Senior fitness test- functional performance-Two Minutes Step Test | baseline and week 12 (after intervention)
  SPPS 29 is validated. In order to perform the test, the participant stands in an upright position; The distance from the front protrusion of the hip bone (iliac crest) to the midpoint of the kneecap (patella) was marked and the midpoint of the distance between these two bones was determined. The participant's step height was determined by marking the height of this determined point from the ground. In order to determine whether the step height reached the target height, a strip was drawn at the determined height or the target height was marked on the wall and it was checked whether the participant's step height (knee height) reached the target height. The participant was made to step where both knees were, reaching the specified height for 2 minutes. At the end of 2 minutes, the total number of right steps taken correctly was recorded.
Muscle Function- Pelvic floor muscles-Superficial electromyography (EMG) | baseline and week 12 (after intervention)
  SPPS 29 is validated.EMG measurement; It was used to record the bioelectrical activity generated by superficial PFM. In the research, NeuroTrac MyoPlus 4 PRO type EMG device was used. Superficial PFM EMG activities were evaluated using disposable, superficial, self-adhesive, silver-silver chloride (Ag/AgCl) electrodes. The diameter of the circular adhesive electrodes was 3.2 cm. The skin area where the superficial electrodes would be attached was cleaned with an alcohol swab to reduce skin impedance. Superficial electrodes were then placed on the muscles parallel to the muscle fibers: superficial PFM- on both sides of the perineal body. The monopolar reference electrode was placed on the right spina iliac anterior superior (SIAS) to eliminate external signals from outside.
Muscle Function- Abdominal muscles-Superficial electromyography (EMG) | baseline and week 12 (after intervention)
  SPPS 29 is validated.EMG measurement; It was used to record the bioelectrical activity generated by superficial PFM. In the research, NeuroTrac MyoPlus 4 PRO type EMG device was used. Superficial PFM EMG activities were evaluated using disposable, superficial, self-adhesive, silver-silver chloride (Ag/AgCl) electrodes. The diameter of the circular adhesive electrodes was 3.2 cm. The skin area where the superficial electrodes would be attached was cleaned with an alcohol swab to reduce skin impedance. Superficial electrodes were then placed on the muscles parallel to the muscle fibers: superficial PFM- on both sides of the perineal body. The monopolar reference electrode was placed on the right spina iliac anterior superior (SIAS) to eliminate external signals from outside.
Fear of falling-Fall Efficacy Scale (FES) | baseline and week 12 (after intervention)
  SPPS 29 is validated.The first version of the Falls Efficacy Scale (FES) was developed by Tinetti and colleagues in the form of 10 questions covering simple daily living activities to evaluate the fear of falling in the elderly population. It enables the detection and evaluation of the activities that cause fear in people. The Fall Activity Scale-International, which is frequently used today, was developed by Yardley et al.by modifying and preserving the 10 items in the original scale and adding 6 new items. According to this index, as the score increases, the fear of falling increases (scale score between 0-100).
hand grip strength | baseline and week 12 (after intervention)
  Jamar hand dynamometer, which is recommended by the American Association of Hand Therapists and has been found to have high validity and reliability in many studies and is therefore considered the gold standard, was used to measure hand grip strength. Measurement of hand grip and finger grip strengths is the standard position recommended by the American Association of Hand Therapists; It was performed in a sitting position, with the shoulder in adduction and neutral rotation, the elbow in 90 degrees of flexion, the forearm in midrotation and supported, and the wrist in neutral. In the test procedure, 3 measurements were made for hand grip strength, with one-minute breaks between each measurement, and the averages in kg were recorded. Measurements are read in lbs (pounds) and kg.
Knee extensor muscle strength | baseline and week 12 (after intervention)
  Assessment of muscle strength was performed with the Lafayette manual-digital muscle testing device (Lafayette Instrument Company, Lafayette, USA). Lafayette brand digital muscle measuring device is a portable device with a digital display LCD screen and 3 interchangeable heads. The device can provide data such as peak power, time to reach peak power, total test time and average force in kg Newton and pounds.The dynamometer was placed distal to the tibia, with the knee in a 65-degree flexion position, and the measurement was made with the command 'push your knee as hard as possible'.
Ankle dorsi-plantar flexion muscle strength | baseline and week 12 (after intervention)
  Assessment of muscle strength was performed with the Lafayette manual-digital muscle testing device (Lafayette Instrument Company, Lafayette, USA). Lafayette brand digital muscle measuring device is a portable device with a digital display LCD screen and 3 interchangeable heads. The device can provide data such as peak power, time to reach peak power, total test time and average force in kg Newton and pounds.
sleep quality (Pitsburg Sleep Quality Index-PSQI) | baseline and week 12 (after intervention)
  PSQI provides a reliable, valid and standardized measurement of sleep quality. The scale consists of a total of 24 questions. The total score is between 0-21. Sleep quality is classified as good (0-4 points) and poor sleep quality (5-21 points). It was stated that the PSQI score, > 5, had a diagnostic sensitivity of 89.6% and a specificity of 86.5% (kappa = 0.75, p ⩽ 0.001) in distinguishing between good and poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Özge ÇELİKER TOSUN, Study Director — Dokuz Eylul University
Locations (1):
- Melda BAŞER SEÇER, Manisa, Yunusemre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data is saved on my hard disk, I can share it if desired.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: three year
Access Criteria: if it is necessary